CLINICAL TRIAL: NCT03158818
Title: Chronic Hepatitis B Virus Infection in Zambia: a Prospective Clinical Cohort Study
Brief Title: Chronic Hepatitis B Virus Infection in Zambia
Acronym: HUTCH
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Tropical Gastroenterology and Nutrition Group (Unknown); Centre for Infectious Disease Research in Zambia (Other)
Responsible Party: Principal Investigator, Michael Vinikoor, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: F151224005
Record Dates: First submitted 2017-05-08; First posted 2017-05-18 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: HBV; Fibrosis, Liver; Cirrhosis, Liver; Alcoholic Hepatitis; Hepatocellular Carcinoma; Hepatitis, Delta
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis, Alcoholic; Carcinoma, Hepatocellular; Hepatitis D | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collected (up to 15 mL) from a vein in the arm for various tests related to HBV and general health at each visit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HBV mono-infected (Standard of Care): 500 patients in Zambia
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — Routine standard of care per Ministry of Health protocol, including blood draws and examinations.

SUMMARY:
Chronic hepatitis B virus infection is a common condition in Zambia. Among Zambian blood donors, up to 8% are chronically infected with HBV. Despite the burden, awareness of HBV is low in Zambia and the Ministry of Health is in early stages of development of guidelines for HBV screening, treatment, and prevention. The purpose of this clinical cohort study is to characterize the clinical features of chronic HBV infection at UTH and describe treatment and care outcomes. The investigators will enroll 500 adults and follow the cohort for up to 5 years to assess short and long-term viral, serologic, and liver outcomes such as cirrhosis and liver cancer.

DETAILED DESCRIPTION:
Viral hepatitis is the #7 cause of death worldwide, yet it has been neglected when compared to other infectious diseases such as HIV/AIDS, tuberculosis, and malaria. Chronic viral hepatitis is caused by hepatitis C virus and hepatitis B virus and these infections are most common in low and middle-income countries, notably Asia and sub-Saharan Africa. In Zambia there are limited data, but from an HIV cohort, the investigators of this study described 10-12% prevalence of chronic HBV. To raise awareness of viral hepatitis in Zambia and to generate local data to guide policymakers, the investigators will recruit 500 adults with chronic HBV infection and follow the cohort in an observational cohort study. In the study patients would be managed according to standards of care and no experimental or investigational drugs would be used. The investigators will carefully describe patient clinical characteristics and among those who receive drug treatment, the investigators will describe the effectiveness of that treatment in reducing liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* HBV-infected, defined as any single positive HBsAg assay

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* HIV-positive

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 500 adults with chronic HBV infection
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in the percentage of patients with HBV viral suppression (Effectiveness of antiviral therapy in HBV-infected patients) | Baseline and after 1 year of treatment
  The percentage of patients with HBV viral suppression.

SECONDARY OUTCOMES:
Proportion of chronic HBV-infected patients with an indication for antiviral treatment. | baseline, after 1 year of treatment, after 2 years of treatment
  Using WHO HBV guidelines, the investigators will determine the proportion of chronic HBV infected patients in the cohort requiring antiviral treatment.
HBV viral control among patients on antiviral treatment | baseline, after 1 year of treatment, after 2 years of treatment
  The percentage of patients with viral control defined as undetectable HBV viral load after 1 and 2 years of treatment.
Serologic, virologic, and hepatic features of chronic HBV infection in Zambia | 0 to month 60
  HBV patients' demographic characteristics at baseline and clinical characteristics at baseline and at 60 months, including alcohol use disorders diagnosed with AUDIT-C, HBV genotypes, HBV viral loads, prevalence of advanced liver disease (based on non-invasive tests), phase of HBV infection (immune tolerant, HBeAg-positive chronic hepatitis, HBeAg-negative chronic hepatitis, and immune control) - based on international guidance.
Proportion with significant liver fibrosis | 0, 12, 24, 36, 48, and 60 months,
  Measure of liver fibrosis using AST-to-platelet ration index (APRI), Fibrosis 4 (FIB-4) and transient elastography.
Incidence and prevalence of hepatocellular carcinoma (HCC) | baseline and after month 60
  The number of new HCC cases (among those without evidence of HCC at baseline) divided by the time in the cohort study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Vinikoor, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Tropical Gastroenterology and Nutrition Group, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Franklin S, Mouliom A, Sinkala E, Kanunga A, Helova A, Dionne-Odom J, Turan JM, Vinikoor M. Hepatitis B virus contact disclosure and testing in Lusaka, Zambia: a mixed-methods study. BMJ Open. 2018 Sep 21;8(9):e022522. doi: 10.1136/bmjopen-2018-022522. PMID 30244215